CLINICAL TRIAL: NCT05689372
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Regulatory Post Marketing Surveillance (rPMS) Study of Ozempic Solution for Injection 1.34mg/ml (Semaglutide) to Evaluate Safety and Effectiveness in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in Korea
Brief Title: Regulatory Post Marketing Surveillance (rPMS) Study of Ozempic (Semaglutide) to Evaluate Safety and Effectiveness in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in Korea
Status: Not yet recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-4666; 1111-1243-9580 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-12-26; First posted 2023-01-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with type 2 diabetes: Participants will be treated with Ozempic (solution for injection 1.34 milligrams per milliliter [mg/ml] (Semaglutide subcutaneous [s.c.]) according to routine clinical practice conditions for 26 weeks. The physician will determine the dose of Ozempic in accordance with the Korean package insert (K-PI).
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will receive Ozempic (solution for injection 1.34 mg/ml (Semaglutide s.c.) according to routine clinical practice conditions for 26 weeks. The physician will determine the dose of Ozempic in accordance with the K-PI.
  Other Names: Ozempic

SUMMARY:
The aim of this study is to assess the safety and effectiveness of Ozempic initiated according to label in adults with Type 2 Diabetes Mellitus (T2DM) under routine clinical practice conditions. Participants will get Ozempic as prescribed by study doctor. The study will last for about 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The decision to initiate treatment with commercially available Ozempic has been made by the participant/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the participant in this study.
* The participant with T2DM is scheduled to start treatment with Ozempic based on the clinical judgment of their treating physician as specified in the approved label in Korea.
* Informed consent is obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male/female age greater than or equal to (>=) 19 years at the time of signing informed consent.

Exclusion Criteria:

* Participants who are or have previously been on Ozempic therapy.
* Known or suspected hypersensitivity to Ozempic, the active substance or any of the excipients.
* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Female patients who is pregnant, breast-feeding or intends to become pregnant and is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by Korea regulation or practice).
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with T2DM will be treated with Ozempic according to routine clinical practice conditions for 26 weeks. The physician will determine the dose of Ozempic in accordance with the K-PI.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number (incidence) of adverse events (AEs) | From baseline (week 0) to 26 weeks
  Measured as count of events.

SECONDARY OUTCOMES:
Number (incidence) of hypoglycaemia level 3 or level 2 according to American Diabetes Association (ADA) guideline 2020 | From baseline (week 0) to 26 weeks
  Measured as count of events. Level 2 refers to glucose less than (<) 54 milligrams per deciliter (mg/dL) (3.0 millimoles per liter [mmol/L]). Level 3 refers to a severe event characterized by altered mental and/or physical status requiring assistance for treatment of hypoglycaemia.
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to 26 weeks
  Measured in percentage.
Participants achieving HbA1c target < 7.0 percent (%) | At 26 weeks
  Measured as count of participants.
Change in fasting blood glucose (FBG)/fasting plasma glucose (FPG) | From baseline (week 0) to 26 weeks
  Measured in milligrams per deciliter (mg/dl).
Change in post prandial blood glucose (PPBG)/post prandial plasma glucose (PPPG) | From baseline (week 0) to 26 weeks
  Measured in mg/dl.
Change in body weight | From baseline (week 0) to 26 weeks
  Measured in kilogram (kg).
Dose of Ozempic | At 26 weeks
  Measured in milligrams per day (mg/day).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com